CLINICAL TRIAL: NCT03281733
Title: Evaluating Gaps in Care of Malnourished Patients on General Medicine Floors in an Acute Care Setting
Brief Title: Evaluating Gaps in Care of Malnourished Patients
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1505016237R001
Record Dates: First submitted 2017-09-06; First posted 2017-09-13 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Malnutrition
Keywords: malnutrition; adult; hospitalized patients; dietitian; communication; discharge; nutrition
MeSH Terms: conditions — Malnutrition; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: As described in detail in the literature, patients identified with malnutrition are at increased risk of poor clinical outcomes. Despite this knowledge, malnourished patients do not always get optimal nutritional management while admitted into a hospital due to what we describe as gaps in care over the course of their admission.

Objective: We hypothesized that the three main gaps in care were poor RDN/MD communication, excessive time spent NPO for procedures/testing, and/or inaccurate/incomplete dietary discharge instructions. The objectives of this study were to determine and to characterize gaps in nutritional care after a malnutrition diagnosis.

Design: This retrospective study involved post-discharge chart reviews of malnourished adult medicine patients admitted to an acute care facility from September 1- November 30, 2014 (n=242).

DETAILED DESCRIPTION:
To assess the prevalence of gaps in care among malnourished adult medicine patients, we conducted a retrospective study of all adult patients (>18 years old) admitted to a medicine unit at NewYork-Presbyterian- Weill Cornell Medical Center from September 1- November 30, 2014 and diagnosed with malnutrition during that admission. Two independent researchers reviewed the medical charts of 242 patients identified through Humedica with either severe or non-severe malnutrition ICD9 codes (262 or 263.0). Each admission/readmission was counted as a separate episode of care. Readmission was defined as those patients readmitted within 3 months of initial admission. Note, we considered defining readmission to be within 30 days of the initial admit date, but the number of participants meeting this criterion in our sample was too small. Patients were excluded if they were admitted to an intensive care unit (ICU) at any point during their stay. Two RDNs reviewed the first 43 charts and inter-reliability was calculated as well as the individual Cohen's kappa for all questions. Reviewers discussed questions with lower agreement in order to avoid future discrepancies.

A gap in communication with medical team was defined as a delay in the approval or implementation of an appropriate nutritional recommendation made by the RDN (i.e. recommendations or pending orders were not verified/ordered within 48 hours). Procedures/testing gap was defined as when a feeding was held in preparation for or related to procedures or testing (i.e. operating room, imaging, swallowing evaluation, etc.). Discharge gap was defined as when the diet order in the discharge instructions given to patients was not consistent with the RDN's recommendations (i.e. RDN recommends an ONS to continue post discharge but discharge orders do not include it).

Fisher's exact and chi-square tests were used to evaluate the following categorical variables: gender, severe versus non-severe malnutrition and malnutrition context. All statistical analysis was performed with Stata/MP 14.1. This study had Institutional Review Board approval.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria will include the following: Adult Patients; Patients diagnosed with Severe or Non-Severe Malnutrition (defined by ICD-9 codes 262 and 263.0); patients covered by a Hospitalist at Weill Cornell while in-patient from September 1, 2014-November 30, 2014

Exclusion Criteria:

* Exclusion Criteria will include the following: Pediatrics; Patients Admission to ICU during their stay; and, Well-Nourished patients defined as not having Malnutrition diagnosis (defined by ICD-9 codes 262 and 263.0)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with Malnutrition between September 1, 2014-November 30, 2014 covered by Medicine Teams
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2015-11-25 (Actual); Primary Completion 2016-06-05 (Actual); Study Completion 2016-11-23 (Actual)

PRIMARY OUTCOMES:
Frequencies of gaps in care of malnourished patients admitted to an adult general medicine service. | September 1- November 30, 2014
  The specific count of gaps in care will be obtained from expert review by two registered dietitians from the charts of 242 malnourished patients. Gaps that met the predetermined study definitions for gaps in care were counted in our analysis. Gaps in care were subcategorized as communication, testing/procedure, and discharge related.Statistical analyses used chi-square and fisher's exact tests to determine statistical differences between the types of gaps in care and to assess if any demographic information led to a higher frequency of gaps in care.

CONTACTS AND LOCATIONS:
Overall Officials: Renuka Gupta, MD, Principal Investigator — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: No
There is no plan